CLINICAL TRIAL: NCT04086199
Title: Discectomy for Lumbar Active Discopathy: Long Term Functional Outcome Comparison Between Anterior and Posterior Approach: A Retrospective Study
Brief Title: Spinal Approach for Lumbar Active Discopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Régional de la Citadelle (Other)
Collaborators: JM Remacle, MD, Head of Neurosurgery Department, CHR Citadelle (Unknown); Vincent Bonhomme, MD, PhD, University Department of Anesthesia and Intensive Care Medicine, CHR Citadelle (Unknown)
Responsible Party: Principal Investigator, Remacle Thibault, MD, Resident in Neurosurgery Department, PhD Student University Of Liege, Belgium, Centre Hospitalier Régional de la Citadelle
Other Study IDs: Th Remacle
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Surgical Injury; Back Pain Lower Back Chronic
MeSH Terms: conditions — Intraoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anterior discectomy: The discectomy is made by an anterior muscle sparring approach (extraperitoneal).
  Interventions: Procedure: Lumbar discectomy
- Posterior discectomy: The discectomy is made by a posterior approach (posterior midline incision).
  Interventions: Procedure: Lumbar discectomy

INTERVENTIONS:
Procedure: Lumbar discectomy — Lumbar discectomy either by an anterior extraperitoneal approach or by a posterior midline approach.

SUMMARY:
The study aims to study the impact on different surgical approaches for lumbar active discopathy. This inflammatory disease of the disc and adjacent vertebral endplates can induce low back pain with inflammatory-like features. Lumbar fusion is proposed to the patient when conservative management is not enough. This fusion can be obtained by an anterior muscle sparring approach or by a posterior muscle decaying approach.

The goal with this single center retrospective study is to identify the surgical approach that offers to the patient the better long term functional outcome. A phone call would allow us to ask patients a few questions:

* Mcnab's criteria
* Roland Morris Disability Questionnaire

The patients medical file review would also allow us to identify:

* the length of hospital stay for the discectomy (in days)
* incidence of Failed Back Surgery Syndrome
* incidence of redo surgeries
* incidence of adjacent level diseases
* incidence of dural tears and eventual complications (meningitis, orthostatic headaches,...)
* incidence of iliac vessels injuries and eventual complications (thrombosis, need for revascularisation,...)

DETAILED DESCRIPTION:
1) The Roland-Morris Disability Questionnaire

When your back hurts, you may find it difficult to do some of the things you normally do.

This list contains sentences that people have used to describe themselves when they have back pain. When you read them, you may find that some stand out because they describe you today.

As you read the list, think of yourself today. When you read a sentence that describes you today, put a tick against it. If the sentence does not describe you, then leave the space blank and go on to the next one. Remember, only tick the sentence if you are sure it describes you today.

1. I stay at home most of the time because of my back.
2. I change position frequently to try and get my back comfortable.
3. I walk more slowly than usual because of my back.
4. Because of my back I am not doing any of the jobs that I usually do around the house.
5. Because of my back, I use a handrail to get upstairs.
6. Because of my back, I lie down to rest more often.
7. Because of my back, I have to hold on to something to get out of an easy chair.
8. Because of my back, I try to get other people to do things for me.
9. I get dressed more slowly then usual because of my back.
10. I only stand for short periods of time because of my back.
11. Because of my back, I try not to bend or kneel down.
12. I find it difficult to get out of a chair because of my back.
13. My back is painful almost all the time.
14. I find it difficult to turn over in bed because of my back.
15. My appetite is not very good because of my back pain.
16. I have trouble putting on my socks (or stockings) because of the pain in my back.
17. I only walk short distances because of my back.
18. I sleep less well because of my back.
19. Because of my back pain, I get dressed with help from someone else.
20. I sit down for most of the day because of my back.
21. I avoid heavy jobs around the house because of my back.
22. Because of my back pain, I am more irritable and bad tempered with people than usual.
23. Because of my back, I go upstairs more slowly than usual.
24. I stay in bed most of the time because of my back.

Note to users:

This questionnaire is taken from: Roland MO, Morris RW. A study of the natural history of back pain. Part 1: Development of a reliable and sensitive measure of disability in low back pain. Spine 1983; 8: 141-144

The score of the RDQ is the total number of items checked - i.e. from a minimum of 0 to a maximum of 24.

It is acceptable to add boxes to indicate where patients should tick each item.

The questionnaire may be adapted for use on-line or by telephone.

2) Modified Macnab Criteria:

Excellent: No pain, No restriction of mobility, Return to normal work and level of activity

Good: Occasional nonradicular pain, Relief of presenting symptoms, Able to return to modified work

Fair: Some improved functional capacity, Still handicapped and/or unemployed

Poor: Continued objective symptoms of root involvement, Additional operative intervention needed at index level irrespective of length of postoperative follow-up

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from lumbar active discopathy (MODIC 1, 2 or 3) with low back pain as dominant symptom and insufficiently relieved by conservative treatments

Exclusion Criteria:

* Irradiated leg pain as dominant symptom
* Acquired symptomatic spinal canal stenosis requiring decompression
* Previous lumbar surgeries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients treated by lumbar discectomy for active discopathy in a single center, CHR Citadelle, by a single surgeon, Dr JM Remacle between 2009 and 2016.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-02 (Estimated); Study Completion 2020-04-02 (Estimated)

PRIMARY OUTCOMES:
Modified Macnab Criteria | At the time of the phone call, up to 11 years after the surgery

SECONDARY OUTCOMES:
The Roland-Morris Disability Questionnaire The Roland-Morris Disability Questionnaire The Roland-Morris Disability Questionnaire The Roland-Morris Disability Questionnaire | At the time of the phone call, up to 11 years after the surgery
Complications related to the surgery | From date of surgery (lumbar discectomy) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
Length of hospital stay for the discectomy surgery | From date of admission in the hospital for the surgery until the date of release from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No